CLINICAL TRIAL: NCT01924312
Title: Early Detection and Prevention of Mild Cognitive Impairment Due to Cerebrovascular Disease
Acronym: MCI/CVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gregory Jicha, 323-5550 (Other)
Responsible Party: Sponsor-Investigator, Gregory Jicha, 323-5550, Gregory A. Jicha, MD, PhD, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01NR141892; 12-0837-F2L (Other: Univeristy of Kentucky)
Record Dates: First submitted 2013-07-02; First posted 2013-08-16 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Cerebrovascular Disease; Mild Cognitive Impairment
Keywords: stroke, dementia, hypertension, diabetes, hyperlipidemia, smoking, obesity
MeSH Terms: conditions — Cerebrovascular Disorders; Cognitive Dysfunction; Stroke; Dementia; Hypertension; Diabetes Mellitus; Hyperlipidemias; Smoking; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Intervention (Placebo Comparator): A placebo cohort of 40 subjects with MCI related to vascular risk factors (MCI-CVD) will be followed longitudinally with cognitive, imaging, blood and optional spinal fluid biomarkers providing insight into the natural disease course of MCI-CVD. This natural history group will serve as the control group for the treatment arm described below.
  Interventions: Behavioral: Heart Health Intervention
- Treatment Group (Experimental): A cohort of 40 subjects with MCI-CVD will be treated with a nursing-based educational program (Heart Health Intervention) including aggressive symptom monitoring and treatment of vascular risks in a 6 visit intervention block over 12 weeks after baseline and thereafter for every 6 months for the study duration of 3 years. These subjects will be followed identically to the subjects in the natural history arm described in the control group above with cognitive testing, imaging, blood, and optional spinal fluid testing.
  Interventions: Behavioral: Heart Health Intervention

INTERVENTIONS:
Behavioral: Heart Health Intervention — A specialty CVD Risk Clinic will focus on education and individualized treatment programs to modify vascular risks in each subject using the methods developed, tested and shown to successfully reduce multiple CVD risk factors in the HeartHealth Program (HRSA grant, 1D1ARH1606, phase I and 2).

SUMMARY:
Vascular risk factors may account for up to 80% of the memory and thinking problems experienced by our aging population today, by far in excess of that caused by Alzheimer's disease. By doing this study, we hope to learn how vascular risk factors cause memory and thinking changes in the elderly, and whether we can prevent memory and thinking changes by reducing these risk factors. Successful completion of project aims will allow an integrated understanding of mild cognitive impairment caused by vascular risks (MCI-CVD) with the potential for tremendous impact on one of the major healthcare crises facing the nation today.

The study will enroll 80 participants with memory and thinking problems (mild cognitive impairment; MCI) and are at risk for stroke and further difficulties with memory and thinking that may eventually lead to disability and a diagnosis of dementia. Each participant will be randomized into one of two groups (40 in each group) and followed over 36 months. One group will be followed to allow us to understand the natural history of memory and thinking impairment, while the other group will receive intensive education and assistance with vascular risk factor (CVD) control.

DETAILED DESCRIPTION:
This is a randomized, controlled study of intensive medical management and educational programming (Heart Health Intervention) for controlling stroke and vascular risks that may impact your thinking and memory (MCI-CVD). This means that if you choose to enroll, it will be determined by chance ( pulling a number from a hat) whether you will receive the study intervention or standard-of-care treatment. One-half of all subjects will be enrolled in the intervention, while the other one half will not. You will have a 50:50 chance of receiving the intervention, like the flip of a coin. You will be in the study for 36 months if you enroll.

Even if you do are not in the study group receiving medical management and educational programs, we will be monitoring your risks for stroke and vascular risks every 6 months and this information will be provided to your primary doctors, potentially resulting in an increased level of care as a result of your participation in this study.

You must have an individual (spouse, friend, or relative), called a "study partner", who is willing to accompany you to all of the study visits or be available by telephone to communicate changes in your health status over the period of this study.

The study visits include checking vital signs (blood pressure, heart rate weight), regular blood testing at 6 month intervals to monitor your vascular risks (blood sugar, cholesterol levels)as well as ensure your safety throughout the study, yearly brain imaging with MRI scans, and optional spinal fluid collection at enrollment and end of study to help us understand brain changes that cannot be measured in blood.

ELIGIBILITY:
Inclusion Criteria:

1. At least 1 of the following vascular risk factors or on treatment for 1 of these conditions determined by the study physicians to be responsible for the mild memory and thinking problems you experience:

   1. poorly controlled hypertension (systolic blood pressure>130mmHg) or prior history of hypertension associated with congestive heart failure (CHF)
   2. poorly controlled cholesterol (LDL > 70 mg/dL or triglycerides > 150 mg/dL)
   3. cardiomyopathy/congestive heart failure with an ejection fraction < 40%
   4. diabetes with fasting glucose > 110 mg/dL or glycosylated hemoglobin(HgbA1c) > 7.0%
   5. homocysteine > 12umol/L
   6. history of stroke or transient ischemic attack (TIA)
   7. tobacco use > 30 pk/yr history
   8. BMI > 30
2. Age > 55 years
3. Memory complaint
4. Montreal Cognitive Assessment (MoCA)score ≤ 26
5. Either, presence of strategic (caudate, thalamus, subcortical white matter lacunar infarcts or mild to moderate small vessel ischemic changes (T2-positive) felt to be sufficient to explain the cognitive decline (in the clinical judgment of the examining physician)
6. English-speaking

Exclusion Criteria:

1. Functional decline due to cognitive impairment, sufficient to meet clinical criteria for dementia
2. Other medical, non-CVD causes of cognitive decline including but not limited to thyroid dysfunction, vitamin B12 deficiency, renal failure with blood urea nitrogen (BUN) > 30 mg/dL, ammonia > 50 mg/dL, other significant electrolyte abnormalities, extreme hypo (< 70 mg/dL) or hyper-glycemia (> 300mg/dL)…ect.
3. Evidence for comorbid, non-vascular neurologic disease on clinical exam or on imaging (i.e. parkinsonism, focal neurologic deficits, amyotrophic lateral sclerosis(ALS), focal brain lesions other than small lacunar infarcts,…)
4. Focal motor, sensory, visual or auditory deficits that would interfere with cognitive assessments or are suggestive of other brain pathology
5. Vision and hearing with or without assistive devices sufficient to complete study protocol including cognitive test procedures

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
California Verbal Learning Test- Delayed Recall | 36 months
  Memory test for a word list after 30 minutes delay will be compared between baseline and end of study visit.
Brain T2 hyperintensity volume on MRI | 36 months
  Magnetic resonance brain imaging will be performed at enrollment and annually to end of study. Change in volumetric measurement of T2 signal hyperintensities(amount of vascular injury)will be determined for the intervention compared to the placebo group

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MOCA) | 36 months
  The MOCA is a brief cognitive screen that will be compared between baseline and end of study for the interventional group compared to the placebo group
Total brain volume | 36 months
  Magnetic resonance imaging of the brain at baseline and end of study will be compared to determine rate of atrophy between the intervention and placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A. Jicha, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No